CLINICAL TRIAL: NCT05765812
Title: A Phase 1/2 Open-label Study of Debio 0123 in Combination With Temozolomide in Adult Participants With Recurrent or Progressive Glioblastoma and of Debio 0123 in Combination With Temozolomide and Radiotherapy in Adult Participants With Newly Diagnosed Glioblastoma
Brief Title: A Study of Debio 0123 in Combination With Temozolomide in Adult Participants With Recurrent or Progressive Glioblastoma and of Debio 0123 in Combination With Temozolomide and Radiotherapy in Adult Participants With Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0123-GBM-105; 2022-502156-31 (EudraCT Number); U1111-1283-6423 (Other: UTN Number (World Health Organization))
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma IDH (Isocitrate Dehydrogenase) Wildtype; Astrocytoma, Grade III
Keywords: WEE1 inhibitor; Glioblastoma, IDH-wildtype, Grade 4, World Health Organization (WHO) 2021; Astrocytoma, IDH-mutant, Grade 3, WHO 2021
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Lymphoma, Follicular | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Parallel assignment applies to the arm groups within Phase 1 of the study. Sequential assignment will apply to Phases 1 and 2 of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 (Dose Escalation): Arm A - Debio 0123 + Temozolomide (Experimental): Participants will receive intermittent Debio 0123, escalating doses along with temozolomide (TMZ) in each 28-day cycle for up to 2 years.
  Interventions: Drug: Debio 0123; Drug: Temozolomide
- Phase 1 (Dose Escalation): Arm B - Debio 0123 + Temozolomide + Radiotherapy (Experimental): Participants will receive intermittent Debio 0123, escalating doses along with TMZ and concomitant administration of radiotherapy (RT) for up to 6 weeks. As per Protocol _V4.0 Arm B has been permanently halted.
  Interventions: Drug: Debio 0123; Drug: Temozolomide; Radiation: Radiotherapy
- Phase 1 (Dose Escalation): Arm C - Debio 0123 + Temozolomide + Radiotherapy (Experimental): Participants will receive intermittent Debio 0123, escalating doses along with TMZ and concomitant administration of radiotherapy (RT) for up to 6 weeks.
  Interventions: Drug: Debio 0123; Drug: Temozolomide; Radiation: Radiotherapy
- Phase 1 (Dose Expansion): Debio 0123 + Temozolomide (Experimental): Participants will receive Debio 0123, escalating doses along with temozolomide (TMZ) in each 28-day cycle for up to 2 years. Participants will receive one of the 2 selected doses for further investigation.
  Interventions: Drug: Debio 0123; Drug: Temozolomide
- Phase 2: Debio 0123 RD + Temozolomide (Experimental): Participants will receive intermittent Debio 0123 RD along with TMZ in each 28-day cycle for up to 2 years.
  Interventions: Drug: Debio 0123; Drug: Temozolomide

INTERVENTIONS:
Drug: Debio 0123 — Administered as capsules.
Drug: Temozolomide — Administered as capsules.
Radiation: Radiotherapy — Administered in accordance with the local clinical practice and applicable Radiation Therapy Oncology Group (RTOG) or the European Organization for Research and Treatment of Cancer (EORTC) guidelines.
  Arms: Phase 1 (Dose Escalation): Arm B - Debio 0123 + Temozolomide + Radiotherapy; Phase 1 (Dose Escalation): Arm C - Debio 0123 + Temozolomide + Radiotherapy

SUMMARY:
The primary purpose of the Phase 1 (Dose Escalation) of this study is to identify the dose-limiting toxicities (DLTs) of Debio 0123 combined with temozolomide (TMZ) (Arm A) and with TMZ and radiotherapy (RT) (Arms B and C) and to characterize the safety and tolerability of these combinations in adult participants with glioblastoma (GBM). Arm B which was previously added to the protocol, has been permanently halted per the safety monitoring committees' decision on the safety findings of this arm.

The primary purpose of Phase 1 (Dose expansion) of the study is to assess the doses studied under Phase 1 (Dose Escalation) Arm A and identify the recommended dose (RD) for further development.

The Phase 2 will start once the RD Phase 1 has been defined. The primary objective of Phase 2 is to assess the efficacy of Debio 0123 at the RD for further development in combination with TMZ, compared to the standard of care (SOC) in adult participants with GBM.

ELIGIBILITY:
Screening Inclusion Criteria for Phase 1 and Phase 2:

* Signed written informed consent approved before undertaking any study-specific procedures.
* Age ≥18 years of age.
* Willing to provide archived or fresh tumor sample, if available. Receipt of tumor sample is not required for the start of study treatment.
* Adequate bone marrow, hepatic, and renal function.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Willing to practice highly effective methods of contraception.
* Life expectancy of at least 3 months in the best judgment of the Investigator.
* Measurable or non-measurable disease as per RANO criteria by gadolinium (Gd)-based contrast-enhanced brain magnetic resonance imaging (MRI).
* Participants receiving corticosteroids must be on a stable or decreasing dose of ≤4 mg daily dexamethasone (or ≤25 mg prednisone) for the 7 days prior to the start of study treatment.
* Participants with seizures must be adequately controlled on a stable regimen of anti-epileptic drugs.

Additional specific inclusion criteria for Phase 1 and Phase 2:

• A maximum of 1 [for Phase 1 (Dose Expansion) and phase 2] or 2 (Phase 1 Arm A) prior treatment lines of which first-line must be treatment with TMZ-based chemoradiotherapy (TMZ concomitantly with RT).

Note: Only 1 prior line of systemic therapy is allowed; combination therapy with TMZ and RT with or without subsequent TMZ maintenance treatment is considered as 1 systemic line. Prior surgery, radiation, or localized delivery of therapeutic agents (i.e., carmustine-containing wafers [GLIADEL®]) for first recurrence is allowed.

* Documented disease recurrence or progression by diagnostic biopsy or Gd-based contrast-enhanced brain MRI as per RANO criteria.
* KPS ≥60.

Additional specific inclusion criteria for Phase 1 Arm A:

* Participants must have one of the following histopathologically proven diagnoses (WHO 2021):
* GBM Isocitrate dehydrogenase (IDH)-wildtype Grade 4 which may include secondary GBMs (i.e., those that progress from low-grade gliomas).
* Astrocytoma, IDH-mutant, Grade 3

Additional specific inclusion criteria for Phase 1 Arm B and C:

* Participants must have a new, histopathologically proven diagnosis of GBM, IDH-wildtype, Grade 4 (based on WHO 2021), which may include secondary GBMs (i.e., those that progress from low-grade gliomas) if the prior treatment included surgery only.
* KPS ≥70.

Additional specific inclusion criteria for Phase 1 dose expansion and Phase 2:

• Participants must have a histopathologically proven diagnosis of GBM, IDH-wildtype Grade 4 WHO 2021

Additional specific exclusion criteria for Phase 1 Arm A • Prior treatment with more than 2 lines of therapy for GBM, IDH-wildtype, Grade 4, or for astrocytoma, IDH-mutant, Grade 3

Additional specific exclusion criteria for Phase 1 and Phase 2

* Known contraindication to undergoing for Gd-based, contrast-enhanced MRI.
* Any anticancer treatment, monoclonal antibodies/biologics, investigational treatment, or RT with curative intent within 28 days prior to starting study treatment.
* Hypersensitivity to Debio 0123, TMZ, dacarbazine, or any of the excipients found in the formulation for Debio 0123 or TMZ.
* Prior exposure to any WEE1 inhibitor.
* History of other malignancies requiring active treatment in the last 2 years prior to the first dose of study treatment except for superficial bladder cancers, adequately treated low-risk prostate cancer under active surveillance, ductal carcinoma in situ or other carcinomas in situ, and non-melanoma skin cancers (basal cell/squamous cell skin cancer) that have been treated with curative intent.
* Left ventricular ejection fraction (LVEF) below 55%.

Additional specific exclusion criteria for Phase 1 Arm B and C:

* Prior radiation, chemotherapy, biological therapy, interstitial brachytherapy, implanted chemotherapy, therapeutics delivered by local injection or convection-enhanced delivery for GBM.
* Prior therapy that would result in an overlap of the radiation fields.

Additional specific exclusion criteria for Phase 1 dose expansion and Phase 2

• Prior treatment with more than 1 line of systemic therapy for GBM, IDH-wildtype, Grade 4 (based on WHO 2021). Combination therapy with TMZ and RT with or without subsequent TMZ maintenance treatment is considered as 1 systemic line.

[Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation): Number of Participants Experiencing Dose-limiting Toxicities (DLTs) | Phase 1: Arm A: Cycle 1 (Cycle=28 days); Arms B and C: Up to approximately 1.8 months
Phase 1 (Dose Escalation): Number of Participants With At Least One Treatment-emergent Adverse Event (TEAE) | Up to 30 days after the end of treatment (Arm A: Up to approximately 26 months and Arms B and C: Up to approximately 3.5 months)
Phase 1 (Dose Escalation): Number of Participants With Clinically Significant Abnormalities in Laboratory, Vital Signs, Electrocardiogram (ECG), and Echocardiogram (ECHO) Parameters | Up to 30 days after the end of treatment (Arm A: Up to approximately 26 months and Arms B and C: Up to approximately 3.5 months)
Phase 1 (Dose Escalation): Change From Baseline in Karnofsky Performance Status (KPS) Score | Until disease progression or end of study (approximately 66 months)
  KPS is an assessment tool for functional impairment. It is a standard way of measuring the ability of participants with cancer to perform ordinary tasks. The KPS scores range from 0 (death) to 100 (no evidence of disease). A higher score means the participant is better able to carry out daily activities.
Phase 1 (Dose Expansion): Number of Participants With At Least One Treatment-emergent Adverse Event (TEAE) | Up to approximately 26 months
Phase 1 (Dose Expansion): Change from Baseline in Tumor Size Assessed by Objective Response (OR) as per Response Assessment in Neuro-oncology (RANO) Criteria | From the start of study treatment until disease progression or end of study (up to approximately 66 months)
Phase 1 (Dose Expansion): Plasma Concentration of Debio 0123 and its Metabolite | Predose and at multiple timepoints up to 6 hours post dose up to Day 15 of Cycle 1 (Cycle=28 days)
Phase 1 (Dose Expansion): Pharmacodynamic(s) PDy, Change from baseline in Phosphorylated Cell Division Cycle (pCDC2) | Predose and 4 to 6 hours post dose on Day 10 of Cycle 1 (Cycle=28 days)
Phase 2: Overall Survival (OS) | From the start of study treatment until death from any cause or end of study (up to approximately 66 months)

SECONDARY OUTCOMES:
Phase 1 (Dose Expansion): OS | From the start of study treatment until death from any cause or end of study (up to approximately 66 months)
Phase 1 (Dose Escalation): Plasma Concentration of Temozolomide | Phase 1: Predose and at multiple timepoints up to 7 hours post dose up to Day 5 of Cycle 1 (Arm A) and up to Day 29 (Arm B and C)
  The PK of temozolomide will be evaluated in plasma.
Phase 1 (Dose Expansion): Number of Participants With Clinically Significant Abnormalities In Laboratory, Vital Signs, ECG, and (ECHO Parameters) | Up to 30 days after the end of treatment (up to approximately 26 months)
Phase 1 (Dose Expansion): Number of Participants With At Least one TEAE | Up to 30 days after the end of treatment (up to approximately 26 months)
Phase 1 (Dose Expansion): Change From Baseline in KPS Score | Until disease progression or end of study (approximately 66 months)
  KPS is an assessment tool for functional impairment. It is a standard way of measuring the ability of participants with cancer to perform ordinary tasks. The KPS scores range from 0 (death) to 100 (no evidence of disease). A higher score means the participant is better able to carry out daily activities.
Phase 2: Change From Baseline in KPS Score | Until disease progression or end of study (approximately 66 months)
  KPS is an assessment tool for functional impairment. It is a standard way of measuring the ability of participants with cancer to perform ordinary tasks. The KPS scores range from 0 (death) to 100 (no evidence of disease). A higher score means the participant is better able to carry out daily activities.
Phase 2: Number of Participants With Clinically Significant Abnormalities in Laboratory, Vital Signs, and ECG Parameters | Up to 30 days after the end of treatment (up to approximately 26 months)
Phase 2: Number of Participants With At Least One TEAE | Up to 30 days after the end of treatment (up to approximately 26 months)
Phases 1 and 2: Plasma Concentration of Debio 0123 and its Metabolite | Phase1(Dose Escalation):Predose, multiple timepoints upto 8hours postdose upto Day 15 of Cycle 1(Arm A) and upto Day 29(Arms B and C);Phase1(Dose expansion)andPhase2: Predose, multiple timepoints upto 4hours postdose upto Day 15 of Cycle1(Cycle=28 days)
  The pharmacokinetics (PK) of Debio-0123 and its metabolite will be evaluated in plasma.
Phases 1 and 2: Percentage of Participants With Best Overall Response (BOR) Assessed As Per Response Assessment in Neuro-oncology (RANO) Criteria | From the start of study treatment until disease progression or end of study (up to approximately 66 months)
Phases 1 and 2: Percentage of Participants with Objective Response (OR) Assessed As Per RANO Criteria | Up to end of study (approximately 66 months)
Phases 1 and 2: Percentage of Participants With Disease Control (DC) Assessed As Per RANO Criteria | From the start of study treatment until disease progression or end of study (up to approximately 66 months)
Phases 1 and 2: Duration of Response (DOR) Assessed As Per RANO Criteria | Up to disease progression or end of study (up to approximately 66 months)
Phases 1 and 2: Progression Free Survival (PFS) Assessed As Per RANO Criteria | From the start of study treatment until disease progression or death or end of study (up to approximately 66 months)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Debiopharm International SA
Locations (17):
- United States (8):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - New York University Langone Medical Center, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Baylor Scott & White Research Institute, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Spain (8):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Clinica Universidad de Navarra (CUN), Madrid
  - South Texas Accelerated Research Therapeutics (START), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universidad de Navarra (CUN), Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Clinico Universitario de Valencia, Valencia
- Universitaetsspital Zuerich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No